CLINICAL TRIAL: NCT02959138
Title: A Phase 1 Open-Label Study to Evaluate the Pharmacokinetics of GS-9876 in Subjects With Impaired Renal Function
Brief Title: Pharmacokinetics of Lanraplenib in Adults With Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-379-1932; 2016-003823-47 (EudraCT Number)
Record Dates: First submitted 2016-11-07; First posted 2016-11-08 (Estimated); Results first posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Inflammatory Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Moderate Renal Impairment (Cohort 1) (Experimental): Participants with moderate renal impairment and matched healthy controls will receive a single dose of lanraplenib
  Interventions: Drug: Lanraplenib.
- Severe Renal Impairment (Adaptive Cohort 2) (Experimental): Participants with severe renal impairment and matched healthy controls will receive a single dose of lanraplenib
  Interventions: Drug: Lanraplenib.
- Mild Renal Impairment (Adaptive Cohort 3) (Experimental): Participants with mild renal impairment and matched healthy controls will receive a single dose of lanraplenib
  Interventions: Drug: Lanraplenib.

INTERVENTIONS:
Drug: Lanraplenib. — 20 mg (2 X 10 mg) tablets administered orally in a fasted state on Day 1
  Other Names: GS-9876

SUMMARY:
The primary objective of this study is to evaluate the pharmacokinetics (PK) of lanraplenib in participants with impaired renal function relative to matched healthy controls. Participants in this study will be enrolled using an adaptive design that includes up to 3 enrolled cohorts. Based on safety and/or PK data in Cohort 1, participants will be enrolled in adaptive Cohorts 2 and/or 3.

ELIGIBILITY:
Key Inclusion Criteria:

All Individuals

* Have the ability to understand and sign a written informed consent form (ICF), which must be obtained prior to initiation of study procedures
* Have a calculated body mass index (BMI) of ≥ 18 kg/m^2 and ≤ 36 kg/m^2 at screening
* Females of childbearing potential must have a negative pregnancy test at screening and clinic admission (Day -1).
* Individuals have not donated blood within 56 days of study entry or plasma within 7 days of study entry and must refrain from blood donation from clinic admission, throughout the study period, and continuing for at least 30 days following the last dose of study drug.
* Have either a normal 12-lead electrocardiogram (ECG) or one with abnormalities that are considered clinically insignificant by the investigator in consultation with the sponsor
* Must, in the opinion of the investigator, be in good health based upon medical history and physical examination, including vital signs

For Individuals with Renal Impairment

* Must have diagnosis of chronic (> 6 months), stable renal impairment with no clinically significant change in renal function status within 90 days prior to study drug administration (Day 1).
* Have a creatinine clearance (CLcr) < 90 mL/min (using the Cockcroft-Gault method) based on serum creatinine and actual body weight as measured at screening.

For Healthy Matched Controlled Individuals (Individuals with Normal Renal Function)

* Have a CLcr ≥ 90 mL/min (using the Cockcroft-Gault method) based on serum creatinine and actual body weight as measured at screening
* Match in age (± 10 years), gender, and body mass index (± 20%, 18 kg/m^2 ≤ BMI ≤ 36 kg/m^2).

Key Exclusion Criteria:

* Be a lactating female
* Have received any investigational compound within 30 days prior to study dosing
* Have current alcohol or substance abuse judged by the investigator to potentially interfere with individual's compliance or individual's safety as judged by the investigator
* Have a positive test result for human immunodeficiency virus type 1 (HIV-1) antibody, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C virus (HCV) antibody
* Have poor venous access that limits phlebotomy

For Individuals with Renal Impairment

* Require or are anticipated to require dialysis within 90 days of study dosing
* Require during the study or have received moderate or strong inhibitors or inducers of cytochrome P450 (CYP) 3A within 2 weeks prior to study drug administration.

For Healthy Matched Controlled Individuals (Individuals with Normal Renal Function)

* Have taken any prescription medications or over-the-counter medications, including herbal products and antacids, within 28 days prior to start of study drug dosing, with the exception of vitamins and/or acetaminophen and/or ibuprofen and/or hormonal contraceptive medications and/or stable hormone replacement therapy in peri- /post-menopausal female

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (6):
- United States (3):
  - Clinical Pharmacology of Miami, Inc. (CPMI), Miami, Florida
  - Omega Research Consultants, LLC, Orlando, Florida
  - Orlando Clinical Research Center, Orlando, Florida
- APEX GmBH, Munich, Germany
- New Zealand (2):
  - Auckland Clinical Studies, Grafton, Auckland
  - Christchurch Clinical Studies Trust, Christchurch

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hsueh CH, Zheng H, Matzkies F, Mozaffarian A, Medzihradsky O, Tarnowski T, Curry N, and Mathias A. Pharmacokinetics and Short-Term Safety of GS-9876, an Oral Spleen Tyrosine Kinase Inhibitor in Subjects with Renal Impairment. American Society for Clinical Pharmacology and Therapeutics 2019; Washington D.C.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in United States, New Zealand, and Germany. The first participant was screened on 21 November 2016. The last study visit occurred on 05 October 2018.
Pre-assignment Details: 75 participants were screened. Participants in adaptive Cohort 3 (Mild renal impairment) were not enrolled following review of safety and pharmacokinetic (PK) data from participants in Cohort 1 (moderate renal impairment).
Groups:
- Moderate Renal Impairment: Participants with moderate renal impairment received a single oral dose of lanraplenib 20 mg (2 x 10 mg tablets) in a fasted state, on Day 1.
- Severe Renal Impairment: Participants with severe renal impairment received a single oral dose of lanraplenib 20 mg (2 x 10 mg tablets) in a fasted state, on Day 1.
- Healthy Control: Matched healthy control participants received a single oral dose of lanraplenib 20 mg (2 x 10 mg tablets) in a fasted state, on Day 1.
Period: Overall Study
Arm/Group | Moderate Renal Impairment | Severe Renal Impairment | Healthy Control
Started | 10 | 10 | 16
Completed | 10 | 9 | 16
Not Completed | 0 | 1 | 0
Not completed — Enrolled but Never Treated | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all enrolled participants who received lanraplenib. Grouping for the analysis was done based on Clcr.
Groups:
- Severe Renal Impairment: Participants with severe renal impairment received a single oral dose of 20 mg (2 x 10 mg tablets) lanraplenib tablets in a fasted state, on Day 1.
- Healthy Control: Matched healthy control participants received a single oral dose of 20 mg (2 x 10 mg tablets) lanraplenib tablets in a fasted state, on Day 1.
- Total: Total of all reporting groups
Arm/Group | Moderate Renal Impairment | Severe Renal Impairment | Healthy Control | Total
Number analyzed (Participants) | 10 | 9 | 16 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (5.5) | 59 (11.6) | 61 (9.4) | 62 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9 | 18
  Male | 5 | 5 | 7 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5 | 10
  Not Hispanic or Latino | 7 | 7 | 11 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0 | 0
  Race: Asian | 0 | 0 | 1 | 1
  Race: Black | 1 | 1 | 2 | 4
  Race: Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 0
  Race: White | 9 | 8 | 12 | 29
  Race: Other | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 2 | 3 | 3 | 8
  United States | 8 | 2 | 8 | 18
  Germany | 0 | 4 | 5 | 9
Estimated Creatinine Clearance (CLcr) [Mean (Standard Deviation); unit: mL/min] — CLcr was estimated using the Cockcroft-Gault (CG) equation for renal function as recommended by the Food and Drug Administration (FDA) and international guidance documents. CG equation:
  For men: CLcr (mL/min) = ([140-age in years] × [body weight in kg])/(72 × serum creatinine in mg/dL) For women: CLcr (mL/min) = 0.85 × ([140-age in years] × [body weight in kg])/(72 × serum creatinine in mg/dL)
  mL/min | 45.3 (11.46) | 23.4 (4.31) | 104.0 (16.21) | 66.5 (37.96)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Parameter: AUClast of Lanraplenib Presented Based on Range of CLcr
Description: AUClast is defined as the concentration of drug from time zero to the last observable concentration. CLcr was estimated using the CG equation for renal function as recommended by the FDA and international guidance documents. CG equation:
  For men: CLcr (mL/min) = ([140-age in years] × [body weight in kg])/(72 × serum creatinine in mg/dL)
  For women: CLcr (mL/min) = 0.85 × ([140-age in years] × [body weight in kg])/(72 × serum creatinine in mg/dL)
  Participants were classified based on estimated CLcr as:
  Moderate renal impairment: CLcr 30-59 mL/min
  Severe renal impairment: CLcr 15-29 mL/min
  Healthy control: CLcr ≥ 90 mL/min
Time Frame: 0 (predose), 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96 and 120 hours postdose on Day 1
Population: PK Analysis Set included all enrolled participants who took study drug, had at least 1 nonmissing postdose concentration value reported by PK lab for corresponding analytes, based on CLcr. Some healthy control participants matched to participants with moderate renal impairment were also used as matches to participants with severe renal impairment.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- Cohort 1: Moderate Renal Impairment: Participants with moderate renal impairment received a single oral dose of lanraplenib 20 mg (2 x 10 mg tablets) in a fasted state, on Day 1.
- Cohort 1: Healthy Control: Matched healthy control participants to moderate renal impairment cohort, received a single oral dose of lanraplenib 20 mg (2 x 10 mg tablets) in a fasted state, on Day 1.
- Cohort 2: Severe Renal Impairment: Participants with severe renal impairment received a single oral dose of lanraplenib 20 mg (2 x 10 mg tablets) in a fasted state, on Day 1.
- Cohort 2: Healthy Control: Matched healthy control participants to severe renal impairment cohort, received a single oral dose of lanraplenib 20 mg (2 x 10 mg tablets) in a fasted state, on Day 1.
Arm/Group | Cohort 1: Moderate Renal Impairment | Cohort 1: Healthy Control | Cohort 2: Severe Renal Impairment | Cohort 2: Healthy Control
Number analyzed (Participants) | 8 | 8 | 9 | 9
h*ng/mL | 2317.8 (813.83) | 2027.4 (424.52) | 2076.3 (812.99) | 1871.6 (519.06)
Statistical Analysis 1: Comparison: Cohort 1: Moderate Renal Impairment vs Cohort 1: Healthy Control; The Estimate statement was used to produce the point estimate and the corresponding 90% confidence interval of the difference in PK parameters of interest on a logarithmic scale; Test type: Other — The test-to-reference ratio (geometric least squares mean (GLSM) ratio) and associated 90% CI were calculated by taking the exponential of the point estimate and the corresponding lower and upper limits, which was consistent with the two 1-sided tests approach; GLSM ratio = 111.68, 90% CI 2-sided [86.94 to 143.47]
Statistical Analysis 2: Comparison: Cohort 2: Severe Renal Impairment vs Cohort 2: Healthy Control; The Estimate statement was used to produce the point estimate and the corresponding 90% CI of the difference in PK parameters of interest on a logarithmic scale; Test type: Other — The test-to-reference ratio GLSM ratio and associated 90% CI were calculated by taking the exponential of the point estimate and the corresponding lower and upper limits, which was consistent with the two 1-sided tests approach; GLSM ratio = 107.04, 90% CI 2-sided [78.47 to 146.02]

2. Primary Outcome: PK Parameter: AUCinf of Lanraplenib Presented Based on Range of CLcr
Description: AUCinf is defined as the concentration of drug extrapolated to infinite time. CLcr was estimated using the CG equation for renal function as recommended by the FDA and international guidance documents. CG equation:
  For men: CLcr (mL/min) = ([140-age in years] × [body weight in kg])/(72 × serum creatinine in mg/dL)
  For women: CLcr (mL/min) = 0.85 × ([140-age in years] × [body weight in kg])/(72 × serum creatinine in mg/dL)
  Participants were classified based on estimated CLcr as:
  Moderate renal impairment: CLcr 30-59 mL/min
  Severe renal impairment: CLcr 15-29 mL/min
  Healthy control: CLcr ≥ 90 mL/min
Time Frame: 0 (predose), 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96 and 120 hours postdose on Day 1
Population: Participants in the PK Analysis Set were analyzed, based on CLcr. Some healthy control participants matched to participants with moderate renal impairment were also used as matches to participants with severe renal impairment.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohort 1: Moderate Renal Impairment | Cohort 1: Healthy Control | Cohort 2: Severe Renal Impairment | Cohort 2: Healthy Control
Number analyzed (Participants) | 8 | 8 | 9 | 9
h*ng/mL | 2478.7 (908.61) | 2153.0 (435.44) | 2223.4 (855.97) | 1994.2 (528.55)
Statistical Analysis 1: Comparison: Cohort 1: Moderate Renal Impairment vs Cohort 1: Healthy Control; [analysis description as in outcome 1, analysis 2]; Test type: Other — [test comment as in outcome 1, analysis 2]; GLSM ratio = 111.92, 90% CI 2-sided [86.92 to 144.12]
Statistical Analysis 2: Comparison: Cohort 2: Severe Renal Impairment vs Cohort 2: Healthy Control; [analysis description as in outcome 1, analysis 2]; Test type: Other — [test comment as in outcome 1, analysis 2]; GLSM ratio = 107.69, 90% CI 2-sided [79.63 to 145.65]

3. Primary Outcome: PK Parameter: Cmax of Lanraplenib Presented Based on Range of CLcr
Description: Cmax is defined as the maximum concentration of drug. CLcr was estimated using the CG equation for renal function as recommended by the FDA and international guidance documents. CG equation:
  For men: CLcr (mL/min) = ([140-age in years] × [body weight in kg])/(72 × serum creatinine in mg/dL)
  For women: CLcr (mL/min) = 0.85 × ([140-age in years] × [body weight in kg])/(72 × serum creatinine in mg/dL)
  Participants were classified based on estimated CLcr as:
  Moderate renal impairment: CLcr 30-59 mL/min
  Severe renal impairment: CLcr 15-29 mL/min
  Healthy control: CLcr ≥ 90 mL/min
Time Frame: 0 (predose), 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96 and 120 hours postdose on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: Moderate Renal Impairment | Cohort 1: Healthy Control | Cohort 2: Severe Renal Impairment | Cohort 2: Healthy Control
Number analyzed (Participants) | 8 | 8 | 9 | 9
ng/mL | 134.4 (35.47) | 131.6 (33.71) | 118.0 (38.97) | 130.5 (30.77)
Statistical Analysis 1: Comparison: Cohort 1: Moderate Renal Impairment vs Cohort 1: Healthy Control; [analysis description as in outcome 1, analysis 2]; Test type: Other — [test comment as in outcome 1, analysis 2]; GLSM ratio = 102.00, 90% CI 2-sided [81.42 to 127.79]
Statistical Analysis 2: Comparison: Cohort 2: Severe Renal Impairment vs Cohort 2: Healthy Control; [analysis description as in outcome 1, analysis 2]; Test type: Other — [test comment as in outcome 1, analysis 2]; GLSM ratio = 87.80, 90% CI 2-sided [68.14 to 113.13]

4. Secondary Outcome: Percentage of Participants Who Experienced Treatment-Emergent Adverse Events
Time Frame: Day 1 up to Day 31
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Groups:
- Moderate Renal Impairment: Participants with moderate renal impairment received a single oral dose of 20 mg lanraplenib tablets in a fasted state, on Day 1.
- Severe Renal Impairment: Participants with severe renal impairment received a single oral dose of 20 mg lanraplenib tablets in a fasted state, on Day 1.
- Healthy Control: Matched healthy control participants received a single oral dose of 20 mg lanraplenib tablets in a fasted state, on Day 1.
Arm/Group | Moderate Renal Impairment | Severe Renal Impairment | Healthy Control
Number analyzed (Participants) | 10 | 9 | 16
percentage of participants | 60.0 | 55.6 | 12.5

5. Secondary Outcome: Percentage of Participants Who Experienced Graded Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were defined as values that increase at least one toxicity grade from baseline. The most severe graded abnormality from all tests was counted for each participant. The criteria used for grading was Common Terminology Criteria for Adverse Events (CTCAE) v 4.03.
Time Frame: Day 1 up to Day 31
Population: Participants in the Safety Analysis Set were analyzed. Grouping for the analysis was done based on CLcr.
Measure: Number; unit: percentage of participants
Arm/Group | Moderate Renal Impairment | Severe Renal Impairment | Healthy Control
Number analyzed (Participants) | 10 | 9 | 16
percentage of participants
  Any Graded Laboratory Abnormality | 80.0 | 100.0 | 81.3
  Grade 3 or above Laboratory Abnormalities | 30.0 | 44.4 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 31
Description: The Safety Analysis Set included all enrolled participants who received lanraplenib. Grouping for the analysis was done based on CLcr.
Arm/Group | Moderate Renal Impairment | Severe Renal Impairment | Healthy Control
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/16
Other Adverse Events (participants affected / at risk) | 6/10 | 5/9 | 2/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Moderate Renal Impairment (N=10) | Severe Renal Impairment (N=9) | Healthy Control (N=16)
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0
Thirst (General disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 1 | 2
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol: Amendment 1 (2017-01-09): https://cdn.clinicaltrials.gov/large-docs/38/NCT02959138/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-13): https://cdn.clinicaltrials.gov/large-docs/38/NCT02959138/SAP_001.pdf